CLINICAL TRIAL: NCT00701545
Title: A Canadian, Multi-center, Prospective, Open-label, Observational, Pharmacovigilance Study to Assess the Safety of Humate-P® Ivr (Infusion Volume Reduced) in Patients Transitioning From Treatment With Currently Available Humate-P®
Brief Title: A Canadian Study to Assess the Safety of Humate-P® Ivr (Infusion Volume Reduced)
Status: Completed | Type: Observational
Sponsor: CSL Behring (Industry)
Responsible Party: Dr David G. Barnes, CSL Behring Canada, Inc.
Other Study IDs: CSLBC-HP-PM-001
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Von Willebrand Disease
Keywords: von Willebrand disease; VWD, Humate-P®; Infusion volume reduced; ivr
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with von Willebrand disease treated with Humate P® ivr in Canada

SUMMARY:
As part of CSL Behring Canada's continued commitment to ensuring the safety of the new low volume preparation of Humate-P®, CSL Behring Canada proposes to conduct a prospective, multi-center structured data collection of routine management of patients with von Willebrand disease treated with Humate P® ivr in Canada. The surveillance will be non-interventional and non-experimental. During the observation period, the routine medical care of the patient will be documented.

It is expected that there will be no difference in the safety and tolerability of Humate-P® ivr compared to Humate-P®

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of any age;
* Patients who are suffering with von Willebrand disease previously treated with Humate-P®;
* Patients who are able to communicate well with the Investigator and his/her representatives;
* Patients who are able and agreeing to comply with all study requirements;
* Patients who have provided written signed and dated informed consent prior to any study procedures being performed.

Exclusion Criteria:

* Patients who have received any investigational drug ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with von Willebrand disease treated with Humate P® ivr in Canada
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2008-02; Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of Humate-P® (reported adverse events) | 6 months

SECONDARY OUTCOMES:
To capture efficacy data on Humate-P® ivr: • supporting clinical management of bleeding episode or surgery • incidence of relevant bleeding episodes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David G. Barnes, Dr., Study Director — CSL Behring Canada
Locations (1):
- Toronto, Canada